CLINICAL TRIAL: NCT01962636
Title: Umbilical Cord Blood Transplantation Using a Myeloablative Preparative Regimen for the Treatment of Hematological Diseases
Brief Title: Umbilical Cord Blood Transplantation Using a Myeloablative Preparative Regimen for Hematological Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013OC013
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Lymphocytic Leukemia (ALL); Chronic Myelogenous Leukemia; Plasma Cell Leukemia; Myelofibrosis; Myelodysplasia; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Marginal Zone B-Cell Lymphoma; Follicular Lymphoma; Lymphoplasmacytic Lymphoma; Mantle-Cell Lymphoma; Prolymphocytic Leukemia; Diffuse Large B Cell Lymphoma; Lymphoblastic Lymphoma; Burkitt's Lymphoma; Non-Hodgkin Lymphoma; Multiple Myeloma
Keywords: Umbilical Cord Transplant; Acute Myeloid Leukemia (AML); Acute Lymphocytic Leukemia (ALL); Chronic Myelogenous Leukemia; Plasma Cell Leukemia; Myelofibrosis; Myelodysplasia; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Marginal Zone B-Cell Lymphoma; Follicular Lymphoma; Lymphoplasmacytic Lymphoma; Mantle-Cell Lymphoma; Prolymphocytic Leukemia; Large Cell Non-Hodgkin Lymphoma; Lymphoblastic Lymphoma; Burkitt's Lymphoma; Non-Hodgkin Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Plasma Cell; Primary Myelofibrosis; Anemia, Refractory, with Excess of Blasts; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Prolymphocytic; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Whole-Body Irradiation; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Umbilical Cord Blood Transplant (Experimental): The myeloablative preparative regimen will consist of cyclophosphamide (CY), fludarabine (FLU) and fractionated total body irradiation (TBI)followed by umbilical cord blood transplant. Immunosuppressive Cyclosporine and Mycophenylate Mofetil (MMF) will be administered pre- and post UCBT.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total Body Irradiation; Drug: Cyclosporine A; Drug: Mycophenylate mofetil; Biological: Umbilical cord blood

INTERVENTIONS:
Drug: Fludarabine — 25 mg/m^2 IV of Fludarabine will be given over 1 hour on days -8, -7, and -6 pre-UCB transplant.
  Other Names: Fludara
Drug: Cyclophosphamide — 60 mg/kg IV of Cyclophosphamide will be given over 2 hours on days -7 and -6 pre-UCB transplant.
  Other Names: Cytoxan
Radiation: Total Body Irradiation — 165 cGy of total body irradiation will be given twice a day on days -4, -3, -2, and -1.
Drug: Cyclosporine A — Cyclosporine A (CSA) will start day -3 and will be administered PO/IV maintaining a trough level between 200 and 400 ng/mL. For adults the initial dose will be 2.5 mg/kg IV over 1 hour every 12 hours. For children < 40 kg the initial dose will be 2.5 mg/kg IV over 1 hour every 8 hours.
  Other Names: CSA
Drug: Mycophenylate mofetil — Mycophenylate mofetil (MMF) 3 gram/day IV/PO for patients who are ≥ 40 kg divided in 2 or 3 doses. Pediatric patient (<40 kilograms) will receive MMF at the dose of 15 mg/kg/dose every 8 hours beginning day -3.
  Other Names: MMF
Biological: Umbilical cord blood — Pre-medications and UCB infusion will be per current institutional policies/guidelines. The infusion of the first UCB unit should begin within 15 minutes, and no later than 30 minutes after arrival on the Unit. If 2 units are used, both cords will be infused within 30-60 minutes of each other as deemed clinically safe by the BMT attending or designee.
  Other Names: UCB

SUMMARY:
This is a treatment guideline for an unrelated umbilical cord blood transplant (UCBT) using a myeloablative preparative regimen for the treatment of hematological diseases, including, but not limited to acute leukemias. The myeloablative preparative regimen will consist of cyclophosphamide (CY), fludarabine (FLU) and fractionated total body irradiation (TBI).

DETAILED DESCRIPTION:
This is a study to collect routine clinical data from UCBT using unrelated single or double UCB units as an alternative, non-HLA-matched stem cell source for patients with hematological diseases.

* data collection from transplant preparative therapy consisting of treatments with chemotherapeutic regimens and total body irradiation.
* data collection from umbilical cord blood selection and infusion.
* data collection from standard supportive disease and transplant related care.

Pre- and post-transplant medication, UCB selection and infusion, supportive care, and follow-up will be according to the current University of Minnesota BMT guidelines.

An average of 18 patients are expected to be treated on this protocol per year.

ELIGIBILITY:
Inclusion Criteria:

* Eligible Disease Status

  * Acute Myeloid Leukemia (AML): high risk CR1 (as evidenced by preceding MDS, high risk cytogenetics, ≥ 2 cycles to obtain CR, erythroblastic or megakaryocytic leukemia; CR2+. All patients must be in CR as defined by hematological recovery, AND <5% blasts by light microscopy within the bone marrow with a cellularity of ≥15%.
  * Very high risk pediatric patients with AML: Patients <21 years, however, are eligible with (M2 marrow) with < 25% blasts in marrow after having failed one or more cycles of chemotherapy.
  * Acute Lymphocytic Leukemia (ALL): high risk CR1 as defined by cytogenetics (such as t(9;22), t (1:19), t(4;11), other MLL rearrangements, hypodiploidy, or IKZF1 abnormalities), DNA index < 0.81, > 1 cycle to obtain CR or presence minimal residual disease (MRD). Patients in CR2+ are eligible. All patients must be in CR as defined by hematological recovery, AND <5% blasts by light microscopy within the bone marrow with a cellularity of ≥15%.
  * Very high risk pediatric patients with ALL: patients <21 years are also considered high risk CR1 if they had M2 or M3 marrow at day 42 from the initiation of induction or M3 marrow at the end of induction. They are eligible once they achieved a complete remission.
  * Chronic Myelogenous Leukemia excluding refractory blast crisis: To be eligible in first chronic phase (CP1) patient must have failed or be intolerant to imatinib mesylate.
  * Plasma Cell Leukemia after initial therapy, who achieved at least a partial remission
  * Advanced Myelofibrosis
  * Myelodysplasia (MDS) IPSS INT-2 or High Risk (i.e. RAEB, RAEBt) or Refractory Anemia with severe pancytopenia or high risk cytogenetics: Blasts must be < 10% by a representative bone marrow aspirate morphology.
  * Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL), Marginal Zone B-Cell Lymphoma or Follicular Lymphoma are eligible if there was disease progression/relapse within 12 of achieving a partial or complete remission. Patients who had remissions lasting > 12 months, are eligible after at least two prior therapies. Patients with bulky disease (nodal mass greater than 5 cm) should be considered for de-bulking chemotherapy before transplant.
  * Lymphoplasmacytic Lymphoma, Mantle-Cell Lymphoma, Prolymphocytic Leukemia are eligible after initial therapy in CR1+ or PR1+.
  * Large Cell NHL > CR2/> PR2: Patients in CR2/PR2 with initial short remission (<6 months) are eligible.
  * Lymphoblastic Lymphoma, Burkitt's Lymphoma, and other high-grade NHL after initial therapy if stage III/IV in CR1/PR1 or after progression if stage I/II < 1 year.
  * Multiple Myeloma beyond PR2: Patients with chromosome 13 abnormalities, first response lasting less than 6 months, or β-2 microglobulin > 3 mg/L, may be considered for this protocol after initial therapy.
  * Myeloproliferative Syndromes
* Availability of suitable UCB unit(s)
* 0 to 55 years
* Voluntary written consent (adult or parental/guardian)

Exclusion Criteria:

* previous irradiation that precludes the safe administration of TBI - Radiation Oncology will evaluate all patients who have had previous radiation therapy
* chemotherapy refractory large cell and high grade NHL (ie progressive disease after > 2 salvage regimens)
* if ≤ 18 years old, prior myeloablative transplant within the last 6 months. If >18 years old prior myeloablative allotransplant or autologous transplant
* extensive prior therapy including > 12 months alkylator therapy or > 6 months alkylator therapy with extensive radiation
* pregnant or breastfeeding
* HIV positive

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-12; Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Survival at 1 year post-transplant | 1 year
  The number of patients that are still living 1 year after UCBT.

SECONDARY OUTCOMES:
Incidence of neutrophil engraftment at day 42. | 42 days
  Number of subjects with neutrophil engraftment at day 42 post UCBT.
Platelet engraftment at 1 year. | 1 year
  Number of patients with platelet engraftment at 1 year post UCBT.
Pattern of chimerism after transplant. | 1 year
  Pattern of chimerism after transplant. Chimerism will be plotted with box-plots and described over time.
Incidence of graft failure. | 100 days
  Cumulative incidence of graft failure after UCBT.
Incidence of acute graft versus host disease at 100 days. | 100 days
  Cumulative incidence will be used to estimate acute graft versus host disease 100 days after UCBT.
Incidence of chronic graft versus host disease at 1 year. | 1 year
  Cumulative incidence will be used to estimate chronic GVHD at 1 year post UCBT.
Incidence of transplant related mortality at 6 months. | 6 months
  Cumulative incidence will be used to estimate transplant related mortality at 6 months post UCBT.
Incidence of disease free survival | 1, 2 years
  Kaplan-Meier curves will be used to estimate disease-free survival at 1 and 2 years post UCBT.
Incidence of overall survival. | 1, 2 years
  Kaplan-Meier curves will be used to estimate overall survival at 1 and 2 years post UCBT.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Brunstein, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota, United States